CLINICAL TRIAL: NCT00647764
Title: Phase 1 Study Of SNX-5422 Mesylate In Adults With Refractory Solid Tumor Malignancies And Lymphomas
Brief Title: Safety Study Of SNX-5422 To Treat Solid Tumor Cancers And Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Esanex Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1311003; PO7318
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Solid Tumor Malignancy; Lymphoid Malignancy (Lymphoma and CLL); Leukemia; Lymphoma
MeSH Terms: conditions — Lymphoma; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: SNX-5422 Mesylate Hsp90 inhibitor

INTERVENTIONS:
Drug: SNX-5422 Mesylate Hsp90 inhibitor — dose escalated, tablets twice a week; undetermined duration until disease progression

SUMMARY:
Hsp90 is a chemical in the body that is involved in promotion of cancer. SNX-5422 is an experimental drug that blocks Hsp90. It is being evaluated for safety and efficacy in patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Solid tumors or lymphoid malignancies refractory to standard therapy
* measurable disease
* recovery to Grade < 1 toxicity due to prior adverse event or chemotherapy
* no chemotherapy within 4 weeks of entering study
* Age > 18 years
* Karnofsy >= 60%
* Life expectancy > 3 months
* normal or adequate organ and marrow function

Exclusion Criteria:

* receiving other investigational agents
* brain metastases
* uncontrolled medical illness
* HIV+ receiving combination antiretroviral therapy
* significant GI disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
MTD, safety and toxicity | continuous

SECONDARY OUTCOMES:
pharmacokinetic profile of SNX-5422 | first cycle
tumor response measured by X-rays or scans | after every 2 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Bethesda, Maryland, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1311003&StudyName=Safety%20Study%20Of%20SNX-5422%20To%20Treat%20Solid%20Tumor%20Cancers%20And%20Lymphomas